CLINICAL TRIAL: NCT05241782
Title: Cathay General Hospital
Brief Title: The Effect of Auricular Acupressure on the Improvement of Anxiousness, Depression and Heart Rate Variability in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cathay General Hospital (Other)
Collaborators: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Hsin-tung Chen, Principal Investigator, Cathay General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CGH-P110017
Record Dates: First submitted 2022-01-26; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Post-stroke Depression; Auricular Acupressure
Keywords: stroke; heart rate variability; autonomic nerve; auricular acupressure; depression; anxiety
MeSH Terms: conditions — Stroke; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group will receive acupressure treatment by the second week, trice daily, 3~5minutes each session for a course of four weeks.
  Interventions: Other: auricular acupressure
- Control group (No Intervention): Experimental group will receive routine care for a course of four weeks.

INTERVENTIONS:
Other: auricular acupressure — Auricular therapy, as defined by Oleson, refers to "a healthcare modality by stimulating the external surface of the ear to alleviate pathological conditions in other parts of the body"Experimental group will receive acupressure treatment by the second week, trice daily, 3~5minutes each session for a course of four weeks
  Arms: Experimental group

SUMMARY:
Heart rate variability (HRV) in post-stroke patients are closely related to patient mortality, neurological deterioration and overall prognosis. Anxiety and depression will demotivate the patients' will to undergo rehabilitation program, which would delay their functional recovery. The influence of acupressure over the auricle on the HRV, anxiousness and depressive mood have yet to be verified. The investigators aimed to study the effect on auricular acupressure treatment between the different trending of HRV, anxiety and depression and their correlations.

This is a randomized control study, consisted of 70 patients with post-stroke depressive mood, from both CGH and Xizhi Cathay hospital in Taiwan. HRV analysis is performed on the first 24 hours, and on a weekly basis for a total of 6 weeks. The included depressed patients were defined by the "Hospital Anxiety and Depression Scale" and weekly will be undertaken by the patients. A "Taiwanese Depression Questionnaire" pre-test and after-test will be undertaken by the patients. Experimental group will receive acupressure treatment by the second week, trice daily, 3~5minutes each session for a course of four weeks. Data were analyzed using SPSS 20.0, using generalized estimating equation, GEE.

The study hypothesized that the auricular acupressure treatment would improve post-stroke depression. Therefore, participants would be more willing to receive rehabilitation program. Our study would also help to provide future references on related studies.

ELIGIBILITY:
Inclusion Criteria:

1. over 20 years old
2. Within 24 hours of arriving at the hospital with the first symptoms of stroke
3. Hemorrhagic stroke:nontraumatic hemorrhagic stroke and Intracerebral Hemorrhage score 0-1
4. Infarct stroke:National Institutes of Health Stroke Scale less than 30
5. Able to express themselves through oral or written communication
6. Hospital Anxiety and Depression Scale Score equal to or greater than 11

Exclusion Criteria:

1. Previous diagnosis of arrhythmia
2. Mental illness, dementia, Alzheimer's disease, or possible complete paralysis on imaging
3. Subarachnoid hemorrhage, subdural hemorrhage, epidural hemorrhage
4. Patients with acute myocardial infarction
5. There is a wound or lesion at the ear auricular point

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-05-14 (Actual); Primary Completion 2022-05-13 (Estimated); Study Completion 2022-08-13 (Estimated)

PRIMARY OUTCOMES:
Taiwanese Depression Questionnaire | 4 Weeks
  The Taiwanese Depression Questionnaire(TDQ), which is a 4-point scale with 18 items, is a culturally specific depression self-rating instrument for effective screening of depression in Taiwan and has satisfactory reliability and validity. Subjects are guided to rate each item on a scale from 0 to 3 on the basis of "how often you felt the physical and emotional aspects during the past week". TDQ scores range from 0 to 54. The original test authors defined three ranges for both of the scales: 0-13 (non-cases), 14-18 (doubtful cases), and 19-54(cases). The higher the score, the more severe the depression.The Taiwanese Depression Questionnaire(TDQ) had a sensitivity of 0.89 and a specificity of 0.92 .
Hospital Anxiety and Depression Scale | 4 Weeks
  The reliability of the HADS was good, with Cronbach's α coefficients of 0.86 (anxiety), 0.85 (depression), and 0.91 (total scale).The HADS consists of 14 items. Seven of the items indicate anxiety and the remaining seven items indicate depression. Each item had been answered by the patient on a four point (0-3) response category so the possible scores ranged from 0 to 21 for anxiety and 0 to 21 for depression.
  The original test authors defined three ranges for both of the scales: 0-7 (non-cases), 8-10 (doubtful cases), and 11-21(cases). It is possible to calculate a HADS total score by simply summing up the anxiety and depression items.

SECONDARY OUTCOMES:
Heart rate variability (HRV) | 4 weeks
  ANSWatch-Mini measures the following physiological parameters while sitting or lying in 6 minutes:Heart rate variability (HRV) HRV is further categorized into frequency bands, the most important of which are the low frequency (LF) and high frequency (HF) components.
  LF and LF/HF ratio were interpreted as indices for sympathetic activation This means HF could be a highly informative biomarker, as it can provide insight into the functional relevance of vagal activity during stress and its role in depression.
  we review relevant studies on HR, HF-HRV and consider their rele vance as markers for clinical groups in the depression-anxiety spectrum for integration to new patient stratification systems.

CONTACTS AND LOCATIONS:
Locations (1):
- Cathay General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided